CLINICAL TRIAL: NCT03635138
Title: Effect of the Incoportation of Copper and Zinc Nanoparticles Into Dental Adhesives on Their Antimicrobial Properties and Dentinal Matrix Metalloproteinases Activity: From Molecular Basis to Clinical Trials
Brief Title: Effect of the Incoportation of Copper and Zinc Nanoparticles Into Dental Adhesives
Acronym: 1170575
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Profesor Titular, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fondecyt 1170575
Record Dates: First submitted 2018-08-06; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Caries, Dental
MeSH Terms: conditions — Dental Caries | interventions — Metal Nanoparticles; Copper; Dental Cements; Nanoparticles

STUDY DESIGN:
Intervention Model Description: Split mouth, 2 premolars restored with 2 dental adhesives , 1 experimental and 1 control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Bottles with a label remarked with 2 letters A and B , same aspect
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adhesives Cu/Zn nanoparticles doped (Experimental): Adhesive dopped with Zn Oxide + Cu nanoparticles in a ( 5% / 0.2% concentration )
  Interventions: Other: Metal nanoparticles ( O Zn and Cu)
- Adhesive control (Active Comparator): Adhesive conventional
  Interventions: Other: Dental Adhesive pure

INTERVENTIONS:
Other: Metal nanoparticles ( O Zn and Cu) — Np of OZn nanoparticles mixed with dental adhesive
  Arms: Adhesives Cu/Zn nanoparticles doped
Other: Dental Adhesive pure — Dental Adhesive with commercial preparation
  Other Names: Dental Adhesive without nanoparticles
  Arms: Adhesive control

SUMMARY:
The hypothesis is that Addition of copper or zinc nanoparticles to a dental adhesive confers antimicrobial and enzymatic degradation-resistant properties, retaining its adhesion mechanical properties and biocompatibility. To corroborate this hypothesis two groups of a dental adhesive doped with copper or zinc nanoparticles should be develop with a respective structural characterization by SEM-EDX, AFM and FTIR. This should be followed by a test of the antimicrobial activity of adhesive and a study of the influence of adhesive nanocomposites on matrix metalloproteases levels and/or activity in vitro to determine some concentrations more relevant. These would proceed to next stage. With the selected adhesive doped concentrations should be evaluate mechanical properties of doped adhesives and assess the biocompatibility by assays in primary cultured gingival fibroblast and cells type odontoblasts. Finally, once the concentration of either Cu- or Zn-doped adhesives is known, these will be evaluated with a clinical design phase in an in vivo model to study antimicrobial properties, matrix metaloproteases levels and/or activity. We will also study biocompatibility of adhesive nanocomposites and mechanical properties to corroborate the in vitro and ex vivo properties determined. There are results using copper nanoparticle on biomaterials that corroborates some properties such as antimicrobial activity against various species and copper release. All the evidence suggests that at low concentrations of copper nanoparticles, there are no significant effects on mechanical properties but with added antibacterial properties on the adhesive

DETAILED DESCRIPTION:
General Objective To evaluate the influence of the incorporation of copper or zinc nanoparticles into a dental adhesive on its antimicrobial action and their influence on dentin matrix metalloproteases activity. To analyze adhesive mechanical properties and biocompatibility Specifics Objectives

1. To develop and structurally characterize a dental adhesive doped with copper or zinc nanoparticles.

   1.1. Preparation of adhesive nanocomposites; 1.2. Structural characterization of adhesive nanocomposites.
2. To assess mechanical, biochemical and functional effects of adhesive nanocomposites in vitro. Assays will be addressed comparing addition of control adhesive, or the adhesive doped with either copper or zinc on fresh recent extracted teeth.(ex vivo phase) 2.1. To test the antimicrobial activity of adhesive; 2. 2. To study the influence of adhesive nanocomposites on matrix metalloproteases levels and/or activity;2.3. To evaluate mechanical properties of adhesive;2.4. To assess biocompatibility. Viability assays in primary cultured gingival fibroblast will be addressed.
3. To evaluate in vivo model (clinical phase) antimicrobial properties, matrix metalloproteases and cathepsin B levels and/or activity, biocompatibility of adhesive nanocomposites in vivo and mechanical properties. Premolars indicated for extraction will be restored using either traditional adhesive or the adhesive nanocomposite. After a month, premolars will be extracted and analyzed as described.

3.1. To determine surface antimicrobial properties of adhesive nanocomposites; 3.2. To assess matrix metalloproteases and cathepsin B levels and/or activity in dentin tissue macerated;3.3 To determine biocompatibility. Dental pulp will be obtained from extracted premolars, and molecular markers of cell viability or cell damage will be addressed of adhesive nanocomposites;3.4 To evaluate mechanical properties of adhesive.

METHODS

1. To develop a dental adhesive doped with copper or zinc nanoparticles. 1.1. Preparation of adhesive nanocomposites (1): CuNP/adhesive nanocomposites will be prepared using the one-bottle adhesive system Prime & Bond 2.1 (Dentsply Caulk, Milford, DE). This acetone-based adhesive contains a mixture of urethane dimethacrylate and acidic monomer dipentaerythritolpentaacrylatemonophosphate. To prepare the adhesive nanocomposites, appropriate amounts of nanoparticle powder (CuNp and ZnNp, Sigma Aldrich, Santiago, Chile) will be weighed and added directly to the adhesive bottle under constant magnetic stirring. The suspension will then be further dispersed in an ultrasonic bath at 37°C for 10 minutes. Adhesive nanocomposites will be prepared with CuNP content in the 0.015 to 0.045 wt.% range according to previous data from our laboratories. The five concentrations of Cu and Zn-doped adhesives will be 0.0150%, 0.0075% and 0.00038% (concentrations with antibacterial active properties based in our previous data (Cu 1-2-3 and Zn 1-2-3).

   1.2. Structural characterization of adhesive nanocomposites (1): Morphology and composition of the nanocomposite adhesive materials will be characterized by SEM-EDX in backscattered electron mode to produce phase contrast and AFM microscopy. The chemical structure of the polymer matrix and residual monomer contents will be analyzed by attenuated total reflection Fourier transform infrared and Raman spectroscopies. The residual monomer will be analyzed considering the carbon-to-carbon double bond vibration of the acrylic monomer in the 1684 - 1636 cm-1 range.
2. To assess antibacterial, mechanical, biochemical and functional effects of adhesive nanocomposites in vitro and ex vivo. Assays will be addressed comparing addition of regular adhesive, or the adhesive doped with either copper or zinc.

   2.1. Assaying antimicrobial properties of adhesive nanocomposite (2) 2.1.1 Antibacterial activity: Briefly, 10-mm discs 2 mm in thickness will be fabricated using resin composite (Filtek Supreme Ultra; 3M, St. Paul, MN) and either left uncoated (control) or coated with the adhesive Prime&Bond 2.1, and equivalent experimental adhesive blends of twelve groups and polymerized according to manufacturers recommendations for 10 seconds using an LED light curing unit (Radii Cal,SDI,AU) at a power density of 1000 mW/cm2. Amalgam discs (Contour; Kerr, Orange, CA) will be fabricated as previously described and used as an additional positive control. A total of fourteen study groups with eight specimens per group will be evaluated in this part of the experiment: (1) control; (2) amalgam (metallic material used like positive control) and 3) Cu 1, 4) Cu 2, 5) Cu 3,6) Zn1,7) Zn2 and 8) Zn3. To ensure removal of unpolymerized monomer, the discs will be immersed in 10 mL sterile deionized water and agitated for 2 hours at 200 rpm and 37.8°C, after which the discs will be left to dry at room temperature for at least 24 hours. The discs will be sterilized by incubation in 70% ethanol for 10 minutes and then aseptically dried for a minimum of 48 hours. The surface of each disc will be inoculated with 100 mL of a defined viable concentration of 1 108 cells/mL anaerobically grown Streptococcus mutans, ATCC1 25175 in brain heart infusion (BHI; 211059; Becton, Dickinson and Company, Franklin Lakes, NJ) broth. To determine the viable cell concentration for each treatment group in colony forming units per mL (CFU/ml), the inoculated discs will be anaerobically after which the total number of recovered CFUs will be determined.

   2.2. In vitro and ex vivo evaluation of MMPs' activity (1-2) 2.2.1 MMP activity inhibition assay (in vitro): Quantitative MMP-2, MMP-8 and MMP-9 activity in vitro will be determined by commercial MMP fluorometric assay kits (SensoLyte assay kits; AnaSpec, San Jose, CA, USA) for screening of the anti-MMP activity. Cu and ZnNP doped adhesives at different concentrations and controls with no Cu or ZnNP adhesives will be added to the reaction buffer, and the assay will be performed according manufacturer's recommendations. Upon cleavage into 2 separate fragments by MMP, the fluorescence of 5-FAM will be monitored by a fluorescent microplate reader (Sinergy TM).

   2.2.2 Determination of MMP activity and levels (ex vivo dentin samples with samples obtained from restored teeth with doped adhesives and control): Twenty-five (n=5) extracted caries-free human third molars will be collected after obtaining patients' informed consent. The teeth will be disinfected in 0.5% chloramine, stored in distilled water, and used within six months of extraction. A small occlusal preparation with standardized dimensions of 3x3x5 mm will be made by a calibrated operator in the center of the tooth using a cylinder diamond bur (109/018, Medium Grit (60730025), Dentsply, NY, USA) and a high-speed hand piece while providing air-water spray. After completing the cavity preparation, it will be filled with resin composite (Filtek Supreme; 3M ESPE). The experimental adhesives doped with Cu and Zn will be used according manufacturer instructions, and the non-doped adhesive will be used as a control on a homologous upper premolar. The resin composite (Filtek Supreme; 3M ESPE) will be applied using the incremental technique. The enamel will be completely removed with a slow-speed diamond saw (Remet, Bologna, Italy) under saline irrigation, and the teeth will be sectioned to obtain 1-mm-thick coronal dentin wafers, which will be subsequently pulverized into powder with a steel hammer. Dentin powder will then be equally divided and demineralized (at 4°C for 24 hrs under stirring) in one of the following water solutions: (1) 0.87 M acetic acid, pH = 2.3; (2) 0.26 M citric acid, pH = 2.3; or (3) 0.5 M EDTA, pH = 6.4; or (4) 0.5 M EGTA, pH = 6.4. Enzyme extraction of the demineralized dentin powder will be suspended in extraction buffer (50 mM Tris-HCl, pH 6.0, containing 5 mM CaCl2, 100 mM NaCl, 0.1% Triton X-100, 0.1% NONIDET P-40, 0.1 mM ZnCl2, 0.02% NaN3) and EDTA-free protease inhibitor cocktail (Sigma Chemical, St. Louis, MO, USA). The samples will then be ultrasonically treated at 40 W output for 3 bursts of 10 secs each at 4°C (Sonicator Ultrasonic Liquid Processor Model W-385, Heat Systems-Ultrasonic Inc., Farmingdale, NY, USA). The vials will be centrifuged at 18,000 rpm for 30 min at 4°C, and the supernatants will be collected. All the proteins present in the supernatants will be precipitated at 4°C by the addition of powdered ammonium sulfate (w/v) to achieve a final concentration of 85% and pH 7.0. The precipitate will be collected by centrifugation at 24,000 rpm for 30 min at 4°C, redissolved in a 10-fold dilution in extraction buffer, dialyzed through a 30-kDa membrane against extraction buffer overnight, and stored at 4°C until analyzed. After this, the dentin powder will be analyzed to assess MMP-2, MMP-9, and cathepsin B activity levels measured by gelatin zymography and to assess MMP-8 by collagen zymography, as previously described.56 Densitometry will be expressed as du (Gel Logic 2200 pro Imaging System, Carestream Health, USA). Briefly, dentin powder samples will be subjected to electrophoresis under non-reducing denaturing conditions in SDS/PAGE gels containing 1 mg/mL of gelatin or 0.1 mg/mL of collagen as substrates. They will then be soaked twice in 2.5% Triton X-100 and incubated for 17 h in developing buffer (20 mM Tris pH 7.4 and 5 mM CaCl2), stained with Coomassie Brilliant Blue R-250, and destained with 10% acetic acid and 20% methanol solution. Levels of MMP-2, MMP-8, MMP-9, cathepsin B, and ICTP (as a marker of dentin collagen hydrolysis) will be determined either by a commercial ELISA Kit or multiplex immunoassays (R&D Systems, Minneapolis, MN, USA, for Luminex technology) according to the manufacturer's recommendations.

   2.3. Mechanical properties testing of adhesive nanocomposites (1-2) Bond strength 2.3.1 Tooth selection and preparation: Seventy extracted caries-free human third molars will be collected after obtaining patients' informed consents of dental clinic of the University of Chile (≈2000 third molar extractions per year, ensuring the availability of these teeth that are normally discarded). The teeth will be disinfected in 0.5% chloramine, stored in distilled water, and used within six months of extraction. A flat dentine surface will be exposed after wet-grinding the occlusal enamel with a #180 SiC paper. The exposed dentine surfaces will be further polished with a wet #600 SiC paper for 60 seconds to standardize the smear layer.

   2.3.2 Experimental design: The teeth will be randomly assigned into twelve groups of five (6 groups per adhesive) , each of which will be treated with a different concentration of doped adhesive .As control without NPs of system Prime & Bond 2.1 (Dentsply Caulk, Milford, DE) will be used.

   2.3.3. Restorative procedure and specimen preparation: The adhesive systems will be applied strictly in accordance with the respective manufacturer's instructions.

   2.3.4 After bonding procedures: All teeth will receive a micro hybrid composite restoration in two increments of 2 mm. Each increment will be light polymerized for 40 seconds using an LED light curing unit at the 1200 mW/cm2 setting (Radii-cal; SDI Limited, Bayswater, Victoria, Australia). Restored teeth will be stored in distilled water at 37°C for 24 hours and then sectioned longitudinally in the mesio-distal and buccal-lingual directions across the bonded interface using a slow-speed diamond saw (Isomet; Buehler Ltd., Lake Bluff, IL) to obtain 15 to 20 resin-dentine sticks, each with a cross sectional area of approximately 0.8 mm2 when measured with a digital caliper (Digimatic Caliper; Mitutoyo, Tokyo, Japan).Each specimen from each tooth will be evaluated for microtensile bond strength (mTBS) except for six randomly-selected resin-dentine bonded specimens, which will be divided for measurement of the in situ degree of conversion (DC) and nanoleakage (NL).

   2.3.5. Microtensile bond strength test: Resin-dentine bonded sticks will be attached to a Geraldeli's jig using cyanoacrylate adhesive and tested under tension (Kratos Dinamometros, Cotia, SP, Brazil) at 0.5 mm/min until failure. The mTBS values will be calculated by dividing the load at failure by the cross-sectional bonding area. The failure mode of the specimens will be classified as cohesive ( failure exclusively within the dentine or resin composite), adhesive (failure at the resin/dentine interface), or mixed (failure at the resin/dentine interface including cohesive failure of the neighboring substrates). Classification will be performed under a stereomicroscope (SZ40; Olympus, Tokyo, Japan) at 100x magnification. Specimens with premature failures (PFs) will be included in the mean.

   2.3.6. Degree of conversion in situ:Three resin-dentine bonded sticks from each tooth will be wet-polished with #1500, #2000, and #2500 SiC paper. They will then be ultrasonically cleaned for 20 minutes and stored in water at 37.8°C for 24 hours before measuring DC. Micro-Raman spectroscopy analysis will be performed using Senterra equipment (Bruker Optik GmbH, Ettlingen, Baden-Wu¨rttemberg, Germany). Calibration of the micro-Raman spectrometer will be performed by resetting it to zero then measuring the coefficient of a silicon specimen. Specimens will be analyzed using the following micro-Raman parameters: 20 mW Neon laser at 532 nm, spatial resolution at 3 mm, spectral resolution at 5 cm-1, accumulation time at 30 seconds with 6 co-additions, and magnification at 110x (Olympus UK, London, UK) to a 1-mm beam diameter. Spectra will be taken at the dentine-adhesive interface at three different sites within the intertubular dentine for each resin-dentine bonded stick. Spectra of unpolymerized adhesives will be used as references. Post-processing of spectra will be performed using the dedicated Opus Spectroscopy Software version 6.5. The ratio of double-bond content of monomer to polymer in the adhesive will be calculated: where ''R'' is the ratio of aliphatic and aromatic peak areas at 1639 cm-1 and 1609 cm-1 in polymerized and unpolymerized adhesives. The in situ DC of all resin-dentine bonded sticks from the same tooth will be averaged for statistical purposes.

   2.3.7. Nanoleakage evaluation: Three resin-bonded sticks from each tooth will be placed in ammoniacal silver nitrate prepared according to the protocol described by Tay et al.57 and stored in darkness for 24 hours. They will then be rinsed thoroughly in distilled water and immersed in photo developing solution for 8 hours under a fluorescent light to reduce silver ions to metallic silver grains within the voids along the bonded interface. Specimens will be wet-polished with a #600, #1000, #1200, #1500, #2000, and #2500 SiC paper and with 1- and 0.25-mm diamond paste (Buehler Ltd., Lake Bluff, IL) using a polishing cloth. They will be ultrasonically cleaned, air dried, mounted on stubs, and coated with carbon-gold (MED 010; Balzers Union, Balzers, Liechtenstein). Resin-dentine interfaces will be analyzed in a field-emission scanning electron microscope operated in the backscattered mode (LEO 435 VP; LEO Electron Microscopy Ltd., Cambridge, UK). Three images will be captured of each resin-dentine bonded stick. The relative percentage of NL within the adhesive and hybrid layers in each specimen will be measured in all images using the Image J software58 by a blinded researcher. Values from the same specimen will be averaged, and the mean NL of all sticks from the same tooth will be average.

   2.4 Assess biocompatibility, viability assays in primary cultured gingival fibroblast 2.4.1 Cell cultures: Primary cultures of human fibroblasts will be obtained by the explant method, from the retromolar tissue of third molars of three male adult individuals.

   Saos-2 human osteosarcoma cell line, commonly used to assess biocompatibility between osteoblast and biomaterials, will be cultured as described by Alcaide et al.60.

   Cells will be seeded in a 96-well plate at a density of 3000 cells per well. After 24h, control culture medium will be replaced by 100 µl of different dilutions of the proper adhesive (10%, 0.1%, 1%, 0.01%, 0%).The plates will be incubated for 24h, 48h and 72h in a 37°C incubator (5%CO2) previous to viability or cell death assays.

   2.4.2 Cell viability and cell cycle analysis: Primary cultures of human fibroblasts will be obtained by the explant method, from the retromolar tissue of third molars of three male adult individuals.

   Saos-2 human osteosarcoma cell line, commonly used to assess biocompatibility between osteoblast and biomaterials, will be cultured as described by Alcaide et al.60.

   Cells will be seeded in a 96-well plate at a density of 3000 cells per well. After 24h, control culture medium will be replaced by 100 µl of different dilutions of the proper adhesive (10%, 0.1%, 1%, 0.01%, 0%).The plates will be incubated for 24h, 48h and 72h in a 37°C incubator (5%CO2) previous to viability or cell death assays.

   2.4.3 Quantitation of viable, early apoptotic, late apoptotic and necrotic cells by fluorescence microscopy: Protocol described by Kasibhatla et al will be used 61. Cells will be stained with an Acridine Orange/Ethidium Bromide solution (AO/EB) and will be examined by fluorescence microscopy. AO will stain both live and dead cells. EB will stain only cells that have lost membrane integrity. Live cells will appear uniformly green. Early apoptotic cells will stain green and contain bright green dots in the nuclei as a consequence of chromatin condensation and nuclear fragmentation. Late apoptotic cells will also incorporate ethidium bromide and therefore stain orange, but, in contrast to necrotic cells, the late apoptotic cells will show condensed and often fragmented nuclei. Necrotic cells stain orange, but have a nuclear morphology resembling that of viable cells, with no condensed chromatin61.

   2.4.4 Detection of apoptosis by phosphatidylserine exposition, DNA laddering and apoptotic mRNA and proteins quantitation: The exposition of phosphatidylserine on the outside surface of the plasma membrane will be analyzed as early signal of apoptosis by staining with annexin V (A5)- allophycocyanin (APC), as described in Alcaide et al60. Fluorescence of the probe APC will be analyzed by flow cytometry.

   The apoptotic DNA ladder assay will be carried out using a DNA ladder Kit (Roche, Germany).

   mRNA and protein levels for tumor suppressor (p53), pro-apoptotic (bax, caspase 3) and anti-apoptotic (bcl-2) mediators will be addressed using quantitative PCR and immunoblot.

   2.4.5 Evaluation of autophagy: To test putative effects of metal NPs on cell autophagy, different autophagy markers will be addressed. Autophagic flux and p62 level will be detected by western blot, and autophagosomes will be visualized by fluorescence microscopy by counting LC3 positive puncta63.
3. Evaluation of metalloprotease levels and/or activity and biocompatibility of adhesive nanocomposites in vivo.

   Premolars indicated for extraction will be restored using either traditional adhesive or the adhesive nanocomposite. After a month (recall by telephonic contact and following the clinic examination), the patients will be examined and premolars will be extracted and analyzed by blinds evaluators (codified by numbers) at all stages as described. Extractions of premolars will be conducted by teachers of dentistry, any effect post-procedure will be assumed and solved by the research team, procedures for patients are free of charge, and everything will be strictly adhered to the recommendations of the ethics committee of the faculty of dentistry of the university of Chile.

   3.1 In vivo evaluation of adhesive nanocomposites: Seventy volunteers who require extraction of the upper right and left first premolars (n = 35 per group) for orthodontic reasons will be selected from the Orthodontic Specialization Program in the clinic of the University of Chile (there will be a recruitment period of 3 months with a co-investigator responsible for monitoring (CB)). Inclusion criteria will be (1) treatment plans indicating premolar extractions for orthodontic reasons, (2) presence of healthy, intact, non-carious, non-restored, and fully erupted treatment teeth, and (3) patients having well-controlled health conditions that allow all procedures to be performed in the research with minimal risk. Exclusion criteria will be (1) patients who do not agree to volunteer for the study and (2) patients not meeting all of the inclusion criteria.A small occlusal preparation will made by a calibrated operator in the center of the tooth using a cylinder diamond bur (.63109/018,Medium Grit (60730025), Dentsply,NY,USA) and a high-speed hand piece while providing air-water spray with standardized dimensions of 3x3x5 mm. After completing the cavity preparation, it will be filled with resin composite (Filtek Supreme; 3M ESPE). The experimental adhesives doped with Cu and Zn will be used according manufacturer instructions, and the non-doped adhesive will be used as a control on the homologous upper premolar and design by simple randomization of parallel groups. The resin composite (Filtek Supreme; 3M ESPE) will be applied using the incremental technique, and finally, one coat of adhesive will be applied as a surface of composite restoration and polymerized for 10 sec. The occlusion will be checked, and the restorations will be finished and polished following manufacturer instructions. Subsequently, polishing and final finishing will used to apply a layer of adhesive on the final restoration, which will be polymerized for 10 seconds (Raddi Cal, SDI, AU). One tooth at a time will be extracted one month after the restorations are made. The patient will receive infiltrative and intraligamental anesthesia (approximately 1.8 mL 2% Mepivacaine (36 mg)) with epinephrine at a ratio of 1:100,000 (18 mg). Then, the teeth will be subjected to tests.

   3.2 Determine surface antimicrobial properties of adhesive nanocomposites: To assess the antibacterial surface properties of doped adhesives, one final layer of adhesives will be applied over the final surface of restorations in a in vivo model. The procedure will be used to assess the number of CFU of S.Mutans on composite surfaces (Main Outcome). Prior to sampling the biofilm, trays will be prepared to print the biofilm over the restorations. For this application, we will use disposable fluoride gel application trays (Deepak Products Inc., Miami, USA), each of which will be sterilized in a biosafety hood (Esco Technologies Inc., Harboro, USA) under ultraviolet light for 30 minutes. Each tray will then be charged with 7.5 ml of TYCSB agar (Casein, yeast extract, L-cysteine, sucrose, bacitracin) (Difco Laboratories Inc., Detroit, MI, USA), which is a selective medium for S. mutans. Subsequently, to individualize the sample collection technique, the trays will be cut to fit no more than 3 teeth. Immediately after this, the trays will be placed in sterile petri plates and stored in sealed plastic bags in a refrigerator. Before use, the trays will be placed in an incubator/stove (ZDP-A2080, LabTech Co., Namyangiu, Korea) for 24 h at 37 °C as a quality control measure. The third and fourth operators will perform the sampling, which will be conducted between 11:00-13:00 to allow for biofilm reorganization following morning brushing. The sampling will be performed by a blind operator gently pressing the tray for 20 s over the RC restoration, followed by homologous RC restoration with and without Cu or Zn-doped adhesive.

   After the sample trays are stored in sterile petri plates, they will be transported at 4 °C and then incubated at 37 °C in a microaerophilic (jar candle CO2 10%) for 48 h. The count of S.mutans will be performed by the fourth operator who will be blinded to the tray was used to print the RC restorations. Later, Gram staining will be performed to determine the micromorphology of the colonies. The S.mutans count will be expressed in colony forming units (CFU) of S.mutans from the plates and trays with the TYCSB agar. Select colonies that will be compatible with S.mutans adhesion and morphological characteristics will be suspended in Todd-Hewitt broth (Difco Laboratories Inc., Detroit, MI, USA) and incubated at 37 °C for 48 h. The colonies will then be subjected to biochemical tests to identify the species of S. mutans and to distinguish it from S. sobrinus. The biochemical tests include raffinose fermentation, melibiose fermentation, and esculin hydrolysis tests. A positive result for all three tests indicates the presence of S. mutans.

   3.3 Assessment of metalloprotease levels and/or activity in macerated dentin tissue will use a similar methodology to that in 2.4.2 3.3.1 Zymography for in situ to assess activities of MMPs 2 and 9 (outcome):A method described by Mazzoni et al.65 will be used on 20 (n=5 per group) freshly extracted non-carious human upper premolars restored by a previous procedure. After removal of the enamel and cementum, 1-mm-thick disks of middle/deep coronal dentin will be obtained. A 1.0-mg/mL stock solution of fluorescein-labeled gelatin was prepared by adding 1.0 mL of water to the vials containing the lyophilized substrate and storing at -20°C until use. The gelatin stock solution is diluted 1:8 with the dilution buffer (NaCl 150 mM, CaCl2 5 mM, Tris-HCl 50 mM, pH 8.0), and an anti-fading agent is added (Mounting Medium with Dapi H-1200, Vectashield, Vector Laboratories LTD, Cambridgeshire, UK). A 50-μL quantity of the fluorescent gelatin mixture is placed on top of each slab and covered with a coverslip. Slides are light-protected and incubated in humidified chambers at 37°C. For identification of the optimum incubation period, fluorescent images are taken from 1 hr to 7 days. Detailed description of the 3D analysis of in situ zymography with confocal microscopy. Briefly, hydrolysis of quenched fluorescein-conjugated gelatin substrate, which is indicative of endogenous gelatinolytic enzyme activity, was assessed by examination under a multi-photon confocal microscope (ex: 488nm, and em: lp530nm; Zeiss, LSM 780, Carl Zeiss, Oberkochen, Germany). Optical sections of 85-μm-thick were acquired from different focal planes, and the stacked images were analyzed, quantified, and processed with ZEN 2010 software (Carl Zeiss).

   3.4. Determination of biocompatibility. Dental pulp will be obtained from extracted premolars, and molecular markers of cell viability (outcomes) or cell damage by adhesive nanocomposites will be addressed.

   Dental pulp will be obtained as described by Vaseemuddin66, from extracted premolars. Total RNA will be separated and mRNA levels of specific apoptosis and autophagy markers will be measured by qPCR, as previously described (2.4.4-2.4.5).

   3.5 Assessment of mechanical properties (nanoleakage and degree conversion analysis to assess the bond stabilities (outcome)) will be equal to methods in 2.1
4. Statistical analysis: Statistical analysis will be performed using SPSS 23.0 software (IBM, New York, NY, USA). Comparisons between quantitative variables (microtensile bond strength, nanoleakage, degree of conversion, count of CFU) between two independent groups will be analyzed by unpaired t test, ANOVA, and pots-hoc test (or respective non-parametric tests according to Shapiro-Wilk testing of data distribution). Associations between sample determinations will be calculated by Pearson's or Spearman's correlation. A power calculation was carried out using data from a previous study67. A sample size with a minimum of 35 patients per group and per each arm of study was needed to find a difference with statistical significance in a CFU final count (main outcome), considering a statistical power of 0.8 based to Vildosola et a study64 (1-β). Significance will be considered if the p value is <0.05. All statistical calculations and their respective powers be corroborated post-hoc according to the data, to determine if it was necessary to increase the sample size in order to improve the statistical power of each comparison, especially for comparison of data obtained from the analysis MMPs activity, considered our primary outcome because in literature there are insufficient data to make a sample calculation a priori.

ELIGIBILITY:
Inclusion Criteria:

1. treatment plans indicating premolar extractions for orthodontic reasons,
2. presence of healthy, intact, non-carious, non-restored, and fully erupted treatment teeth,
3. patients having well-controlled health conditions that allow all procedures to be performed in the research with minimal risk

Exclusion Criteria:

1. patients who do not agree to volunteer for the study
2. patients not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
To assess antibacterial ( by inhibition of UFC grow of S Mutans count) and Micro tensile bond strengh ( | baseline - 1 month post restorative procedure
  UFC (Colony Forming Units) of Stretococus Mutans Count (Numbers) , Microtensile bond strength (Mpa)
In vitro and ex vivo evaluation of MMPs' activity ( Units of fluorecense by inmunofloresence antibody compared with control ) | baseline - 1 month post restorative procedure
  To Assess Matrix Metallopeptidase 2 , 8 and 9 activity by in vitro test and ex vivo (Luminicense units compared vs controls of fluorecence) ( dentin powder obtained fron teeth donated)

CONTACTS AND LOCATIONS:
Locations (1):
- Eduardo Fernández G, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No